CLINICAL TRIAL: NCT05397301
Title: Comparison of Controlled Sedoanalgesia and General Anesthesia in Dacryocystorhinostomy Surgery
Brief Title: Controlled Sedoanalgesia in External DCR Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turkish Society of Anesthesiology and Reanimation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: uludaganesthesia
Record Dates: First submitted 2022-05-22; First posted 2022-05-31 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Dacryocystorhinostomy; Sedation; General Anesthesia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sedoanalgesia(SA group) (Active Comparator): Sedoanalgesia was applied to the SA group
  Interventions: Procedure: Controlled sedoanalgesia
- general anaesthesia (GA group) (Active Comparator): General anaesthesia was applied to the GA group
  Interventions: Procedure: Controlled sedoanalgesia

INTERVENTIONS:
Procedure: Controlled sedoanalgesia — Controlled sedoanalgesia was applied with Bispectral index and dexmedetomidine

SUMMARY:
In our study, we aim to compare general anesthesia and controlled sedoanalgesia methods in dacryocystorhinostomy (DCR) surgery in terms of hemodynamic data, bleeding amount, postoperative complications (bleeding, pain, etc.) and anesthesia satisfaction in a prospective and randomized controlled manner.

DETAILED DESCRIPTION:
The patients were routinely monitored in the operating room in accordance with the standard protocol for elective surgeries, and the preoperative findings (blood pressure, oxygen saturation, cardiac rhythm, peak heart rate) were recorded.

The decision of routine anesthesia was not interfered with. The data of the patients were collected as GA group if general anesthesia was applied and SA group if sedoanalgesia was applied. If general anesthesia was preferred, anesthesia induction was performed with propofol, fentanyl and rocuronium, and sevoflurane was used for anesthesia maintenance. Intravenous midazolam and dexmedetomidine infusions were administered to patients for whom sedoanalgesia was preferred. The sedation level of these patients was followed up with the Ramsay sedation scale (RSS) and capnography monitoring was performed.

Whether general anesthesia or sedoanalgesia was preferred, local anesthesia was administered to all patients by the surgical team and intraoperative hemodynamic data (mean arterial pressure, heart rate, oxygen saturation) were followed.

In addition to patients recruited for the study, hemodynamic data after induction, endotracheal intubation, surgical incision, and extubation were also recorded.

Depth of anesthesia was monitored with a bispectral index monitor for both groups.

Intraoperative bleeding amount, canal damage, etc. Intraoperative complications such as In this study, the pain levels of the patients were evaluated by visual pain score (VAS) at 0 and 30 minutes, 1st, 4th, 8th and 12th hours. Analgesic requirement, postoperative nausea-vomiting and time, duration of surgery, length of hospital stay, surgery-related complications (ecchymosis, epistaxis, hematoma, edema, etc.) were recorded. Patient and surgical team satisfaction of the patients was evaluated using a 5-point Likert Scale.

The necessary measurements of the eyes and adnexa (visual acuity, meibomian gland measurement, tear breakout time, schirmer) for which detailed eye examinations of the patients will be performed preoperatively and postoperatively on the 1st day, 1st week, 1st month, 3rd month and 6th month. tests, intraocular pressure, pupil width, lens density, corneal topography, anterior and posterior segment Optical coherence tomography, etc.) tear duct examination and lavage were performed. The patient's complaints about eye diseases were recorded. As a result of the study, in addition to local anesthesia in DCR surgery, sedoanalgesia and general anesthesia methods were compared.

ELIGIBILITY:
Inclusion Criteria:

* Primary DCR surgery to be performed
* 18 years and older patients
* Having an American Society of Anesthesiology score of 1, 2, 3
* Having approved and signed the informed consent form

Exclusion Criteria:

* Patients younger than 18 years old
* Patients with an American Society of Anesthesiology score of 4 and above
* Patients who do not accept informed consent
* History of drug allergy and opioid tolerance
* Uncontrolled diabetes mellitus
* Coagulation disorder
* Cases with severe liver and kidney disease
* Those who refused to participate in the study
* They will have DCR surgery again

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-02-07 (Actual); Primary Completion 2021-02-07 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
hemodynamic data | through surgery completion
  blood pressure (mm/hg)
hemodynamic data | through surgery completion
  heart rate (bpm)
hemodynamic data | through surgery completion
  peripheral oxygen saturation (percent)
amount of bleeding | amount of bleeding calculated during surgery
  the amount that bleeds into the aspirator and cottons during the surgery (ml)

SECONDARY OUTCOMES:
postoperative complications | postoperatif 12 hour
  pain
postoperative complications | postoperatif 12 hour
  nause and vomiting

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Uludağ Üniversitesi Tip Fakültesi, Bursa, Ni̇lüfer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ciftci F, Pocan S, Karadayi K, Gulecek O. Local versus general anesthesia for external dacryocystorhinostomy in young patients. Ophthalmic Plast Reconstr Surg. 2005 May;21(3):201-6. doi: 10.1097/01.iop.0000163317.73873.c9. PMID 15942495
- [Background] Tuladhar S, Adhikari S, Bhattarai BK. Effectiveness of sedation in dacryocystorhinostomy surgery. Nepal J Ophthalmol. 2009 Jan-Jun;1(1):25-31. doi: 10.3126/nepjoph.v1i1.3670. PMID 21141018
- [Background] Scawn RL, Allen MJ, Rose GE, Verity DH. Randomised, masked study of local anaesthesia administered prior to external dacryocystorhinostomy under general anaesthesia. Eye (Lond). 2019 Mar;33(3):374-379. doi: 10.1038/s41433-018-0201-5. Epub 2018 Sep 18. PMID 30228368
- [Background] Eghbal MH, Sahmeddini MA. Comparison larygeal mask airway with the endotracheal tube for the external dacryocystorhionostomy surgery. A randomized clinical trial. Middle East J Anaesthesiol. 2013 Oct;22(3):283-8. PMID 24649784
- [Background] Kersey JP, Sleep T, Hodgkins PR. Ocular perforation associated with local anaesthetic for dacryocystorhinostomy. Eye (Lond). 2001 Oct;15(Pt 5):671-2. doi: 10.1038/eye.2001.213. No abstract available. PMID 11702990
- [Background] Apan A, Doganci N, Ergan A, Buyukkocak U. Bispectral index-guided intraoperative sedation with dexmedetomidine and midazolam infusion in outpatient cataract surgery. Minerva Anestesiol. 2009 May;75(5):239-44. Epub 2008 Dec 17. PMID 19088698
- [Background] Harissi-Dagher M, Boulos P, Hardy I, Guay J. Comparison of anesthetic and surgical outcomes of dacryocystorhinostomy using loco-regional versus general anesthesia. Digit J Ophthalmol. 2008 Jan 1;14:1-6. doi: 10.5693/djo.01.2008.001. eCollection 2008. PMID 29440968
- [Derived] Saglam U, Kivanc SA, Girgin NK. Comparison of Anesthetic and Surgical Outcomes Between General Anesthesia and Dexmedetomidine-Based Sedoanalgesia in Dacryocystorhinostomy Surgery With Bispectral Index Monitoring. Anesthesiol Res Pract. 2025 Nov 4;2025:6650312. doi: 10.1155/anrp/6650312. eCollection 2025. PMID 41200122